CLINICAL TRIAL: NCT02378597
Title: Developing a Resiliency Program for Medical Interpreters in Cancer Care
Brief Title: Resiliency Program for Medical Interpreters
Acronym: CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Elyse Park, PhD, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-524
Record Dates: First submitted 2014-06-27; First posted 2015-03-04 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Psychological Stress
Keywords: Resiliency burnout stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed Intervention: Control (Active Comparator): Delayed intervention: Control was a a behavioral treatment for resiliency delivered in a single 4 hour session delivered in a delayed fashion (waitlist control)
  Interventions: Behavioral: Behavioral: Resiliency Intervention
- Experimental: Intervention (Experimental): Experimental: Intervention was a 4 hour behavioral resiliency intervention.
  Interventions: Behavioral: Behavioral: Resiliency Intervention

INTERVENTIONS:
Behavioral: Behavioral: Resiliency Intervention — 4 hour behavioral session including education in the relaxation response, education about stress and allostatic load, cognitive skills building, review of difficult encounters with patients.
  Other Names: CARE

SUMMARY:
To develop and test a 4-session program to teach resiliency skills to Medical Interpreters.

DETAILED DESCRIPTION:
This study aims to improve quality of cancer care for LEP patients through improving medical interpreters' ability to cope with difficult encounters. We propose to (1) identify the needs of medical interpreters working with cancer patients, and (2) develop and test a psychoeducational resiliency program at 3 DF/HCC cancer centers: MGH, DFCI, and BWH) intended to enhance interpreters' skills to effectively manage stressful encounters and to cope with the personal effects of encounters.

ELIGIBILITY:
Inclusion Criteria:

1. Interpreter employed at one of the 3 study hospitals
2. >=20 hours/week

Exclusion Criteria:

1) Interpreter working <20 hours per week

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Feasibility and Acceptability of Intervention (participant feedback questionnaire) | Post-Intervention (4 weeks)
  A participant feedback questionnaire will be completed by participants, including questions about whether the logistics and content of the intervention were feasible and acceptable to them. Attendance to the sessions is also considered as a component of feasibility.

SECONDARY OUTCOMES:
Psychological Variables including Perceived Stress and Resiliency ( PSS-1021 is a 10-item scale) | Baseline, Post-Intervention (4 weeks), and 12 week follow up
  The PSS-1021 is a 10-item scale designed to measure the degree to which situations in one's life are appraised, or considered as stressful, and how unpredictable, uncontrollable, and overloaded respondents find their lives. Responses are on 4-item Likert scales and range from 10-40; higher score = greater stress.The Resiliency Scale is a 14-item self-report measure to assess one's ability to successfully deal with adversity.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Russell-Einhorn, JD, Study Director — Dana-Farber Cancer Institute